CLINICAL TRIAL: NCT04971252
Title: Impact of Type II Diabetes Mellitus on Basic Coagulation Profile and Platelet Indices in Non-dialysis Chronic Kidney Disease Patients
Brief Title: Type 2 Diabetes Mellitus and Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Khalaf Mohamed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-21-07-24
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Renal Disorder Associated With Type II Diabetes Mellitus
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — Blood samples for coagulation profile and platelet indices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Co existance of diabetes mellitus and chronic kidney disease: Study basic coagulation profile and platelet indices among those patients with combined diabetes mellitus and chronic kidney disease
  Interventions: Diagnostic Test: Hematologic tests for patients with diabetes mellitus and chronic kidney disease
- Diabetes mellitus without chronic kidney disease: Study basic coagulation profile and platelet indices among those patients with diabetes mellitus only
  Interventions: Diagnostic Test: Hematologic tests for patients with diabetes mellitus and chronic kidney disease
- Chronic kidney disease without diabetes mellitus: Study basic coagulation profile and platelet indices among those patients with chronic kidney disease without diabetes mellitus
  Interventions: Diagnostic Test: Hematologic tests for patients with diabetes mellitus and chronic kidney disease

INTERVENTIONS:
Diagnostic Test: Hematologic tests for patients with diabetes mellitus and chronic kidney disease — Study basic coagulation profile and platelet indices among diabetic patients with chronic kidney disease

SUMMARY:
To investigate the effect of co existance of diabetes mellitus and chronic kidney disease on basic coagulation profile in comparison with diabetic patients with normal kidney function and non diabetic patients with chronic kidney disease

DETAILED DESCRIPTION:
We will study impact of type 2 diabetes mellitus on basic coagulation profile and platelet indices among patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus with and without chronic kidney disease Patients with chronic kidney disease without diabetes mellitus

Exclusion Criteria:

* any situation influence on basic coagulation profile and platelet indices other than diabetes mellitus and chronic kidney disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will classify study population into 3 groups First group those population with only type 2 diabetes mellitus Second group is those population with chronic kidney disease only Third group is those population with combined type 2 diabetes mellitus and chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Estimate risk of thrombosis or bleeding for the 3 study groups by prothrombin time | 1 day
  We will include 150 patients and classify them into 3 groups each one consists of 50 patients First group those patients with diabetes mellitus only Second group those patients with chronic kidney disease only Third group those patients with combined diabetes mellitus type 2 and chronic kidney disease not on hemodialysis First we will measure prothrombin time
Estimate risk of thrombosis or bleeding for the 3 study groups by prothrombin concentration | 1 day
  We will include 150 patients classified into 3 groups as previous Second measure is prothrombin concentration
Estimate risk of thrombosis or bleeding for the 3 study groups by INR | 1 day
  We will include 150 patients as previous Third measure is INR ( international normalised ratio )
Estimate risk of thrombosis or bleeding for the 3 study groups by partial thromboplastin time | 1 day
  We will include 150 patients as previous Fourth measure is partial thromboplastin time
Estimate risk of thrombosis or bleeding for the 3 study groups by serum fibrinogen | 1 day
  We will include 150 patients as previous Fifth measure is serum fibrinogen level in the 3 groups
Estimate risk of thrombosis or bleeding for the 3 study groups by mean platelet volume | 1 day
  We will include 150 patients as previous Sixth measure is mean platelet volume in the 3 groups
Estimate risk of thrombosis or bleeding for the 3 study groups by platelet distribution width | 1 day
  We will include 150 patients as previous Seventh measure is platelet distribution width for the 3 groups
Estimate risk of thrombosis or bleeding for the 3 study groups by plateletcrit | 1 day
  We will include 150 patients as previous Eighth measure is plateletcrit of the 3 study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Gundogan K, Bayram F, Capak M, Tanriverdi F, Karaman A, Ozturk A, Altunbas H, Gokce C, Kalkan A, Yazici C. Prevalence of metabolic syndrome in the Mediterranean region of Turkey: evaluation of hypertension, diabetes mellitus, obesity, and dyslipidemia. Metab Syndr Relat Disord. 2009 Oct;7(5):427-34. doi: 10.1089/met.2008.0068. PMID 19754305
- [Background] Odegaard AO, Jacobs DR Jr, Sanchez OA, Goff DC Jr, Reiner AP, Gross MD. Oxidative stress, inflammation, endothelial dysfunction and incidence of type 2 diabetes. Cardiovasc Diabetol. 2016 Mar 24;15:51. doi: 10.1186/s12933-016-0369-6. PMID 27013319
- [Background] Ulutas KT, Dokuyucu R, Sefil F, Yengil E, Sumbul AT, Rizaoglu H, Ustun I, Yula E, Sabuncu T, Gokce C. Evaluation of mean platelet volume in patients with type 2 diabetes mellitus and blood glucose regulation: a marker for atherosclerosis? Int J Clin Exp Med. 2014 Apr 15;7(4):955-61. eCollection 2014. PMID 24955167